CLINICAL TRIAL: NCT00151814
Title: An Open-label Study of the Single-dose Pharmacokinetics of Olmesartan Medoxomil in Pediatric Patients With Hypertension
Brief Title: Olmesartan Pediatric Pharmacokinetic (PK) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Michael Melino, PhD, Daiichi Sankyo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS0866-A-U102
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Results first posted 2010-04-09 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Hypertension
Keywords: Olmesartan PK in children
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil

ARMS (1):
- Olmesartan (Experimental): Children less than 6 years old received 0.3 mg/kg. Children 6 years old or older received 40 mg, if they weighed 35 kg or more; 20 mg if they weighed less than 35 kg.
  Interventions: Drug: Olmesartan medoxomil

INTERVENTIONS:
Drug: Olmesartan medoxomil — Children less than 6 years old: oral suspension or tablets equal to 0.3 mg/kg; 20 mg or 40 mg tablets for older children depending on weight.

SUMMARY:
Determine single dose pharmacokinetic parameters of olmesartan in pediatric patients with hypertension in ages 12 months - 16 years

ELIGIBILITY:
Inclusion Criteria:

* Age 12 months to 16 years inclusive
* Signed parental/guardian informed consent and assent from the subject
* Current treatment for hypertension, or, if not currently treated for hypertension, systolic blood pressure (SBP) greater than or equal to 95th percentile for gender and height-for-age, or, if not currently treated for hypertension, systolic blood pressure or diastolic blood pressure greater than or equal to 90th percentile for gender and height-for-age and diabetic or having a family history of hypertension
* Glomerular filtration rate (GFR) greater than or equal to 30 mL/min/1.73 m2, estimated using the Schwartz equation
* Sexually active females of child-bearing potential must be practicing an acceptable method of birth control
* Negative serum beta-human chorionic gonadotropin at screening and at admission (female of child-bearing potential only)

Exclusion Criteria:

* Clinically significant cardiac, gastrointestinal, hematologic, hepatic or hepatobiliary, neurologic, or pulmonary (except asthma) disorder
* History of severe or symptomatic hypertension associated with stroke, seizures, encephalopathy, or other significant neurologic findings within 1 year prior to screening
* Current treatment with more than 2 antihypertensive medications
* Secondary hypertension from uncorrected coarctation of the aorta, bilateral renal artery stenosis, or unilateral renal artery stenosis in a single kidney
* Serum albumin < 2.5 g/dL
* Major organ or bone marrow transplantation except for prior kidney transplantation of at least 6 months and with stable renal function meeting the inclusion criteria

Ages: 12 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Little Rock, Arkansas
  - La Jolla, California
  - Louisville, Kentucky
  - Kansas City, Missouri
  - Cleveland, Ohio

REFERENCES:
- [Derived] Wells TG, Blowey DL, Sullivan JE, Blumer J, Sherbotie JR, Song S, Rohatagi S, Heyrman R, Salazar DE. Pharmacokinetics of olmesartan medoxomil in pediatric patients with hypertension. Paediatr Drugs. 2012 Dec 1;14(6):401-9. doi: 10.2165/11631450-000000000-00000. PMID 22880942

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from September 2005 to February 2008. This period lasted for this length of time because of difficulties in recruiting participants. Children from 12 months old to 16 years old were to be enrolled.
Pre-assignment Details: The 2-5 years old cohort had only 4 participants and their data were not sufficient for meaningful analysis. No participants in the 12-23 month old category were enrolled.
Groups:
- Olmesartan Group - 2 to 5 Years Old; Olmesartan Group - 6 to 12 Years Old; Olmesartan Group - 13 to 16 Years Old: Hypertensive children and adolescents of both genders between the ages of 2 years and 16 years of age. The dose for children <6 years old was 0.3 mg.kg; the dose for children > or = to 6 years of age and > or = to 35 kg was 40mg; for <35 kg the dose was 20 mg.
Period: Overall Study
Arm/Group | Olmesartan Group - 2 to 5 Years Old | Olmesartan Group - 6 to 12 Years Old | Olmesartan Group - 13 to 16 Years Old
Started | 4 | 10 | 10
Completed | 4 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olmesartan Group - 2 to 5 Years Old | Olmesartan Group - 6 to 12 Years Old | Olmesartan Group - 13 to 16 Years Old | Total
Number analyzed (Participants) | 4 | 10 | 10 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 4.8 (0.50) | 10.2 (1.03) | 14.8 (1.03) | 11.2 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 5 | 13
  Male | 1 | 5 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 4 | 10 | 10 | 24
Height [Mean (Standard Deviation); unit: cm] | 116.7 (9.01) | 151.8 (9.44) | 165.5 (9.74) | 151.6 (19.44)
Weight [Mean (Standard Deviation); unit: kg] | 32.0 (16.31) | 70.3 (20.53) | 86.3 (29.50) | 70.6 (30.09)

OUTCOME MEASURES:

1. Primary Outcome: For Olmesartan, the Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC 0-t)
Time Frame: PK samples were collected pre-dose and at 1,2,4,8,12,24,48 hours after dosing
Population: 24 participants were enrolled; however, the data for the four 2-5 years old participants were not analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Groups:
- 6-12 Years of Age Olmesartan Group; 13-16 Years of Age Olmesartan Group: Hypertensive children and adolescents of both genders between the ages of 2 years and 16 years of age. The dose for children <6 years old was 0.3 mg.kg; the dose for children > or = to 6 years of age and > or = to 35 kg was 40mg; for <35 kg the dose was 20 mg.
Arm/Group | 6-12 Years of Age Olmesartan Group | 13-16 Years of Age Olmesartan Group
Number analyzed (Participants) | 10 | 10
ng/mL*hr | 7874 (2913) | 5851 (2083)

2. Primary Outcome: For Olmesartan, Area Under the Concentration-time Curve From the Time of the Dose to Infinity
Time Frame: PK samples were collected pre-dose and at 1,2,4,8,12,24,48 hours after dosing
Population: 24 participants were enrolled; however, the data for the four 2-5 years old participants were not analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL*hr
Arm/Group | 6-12 Years of Age Olmesartan Group | 13-16 Years of Age Olmesartan Group
Number analyzed (Participants) | 10 | 10
ng/mL*hr | 7988 (2913) | 5982 (2130)

3. Primary Outcome: For Olmesartan, the Elimination Constant Rate
Time Frame: PK samples were collected pre-dose and at 1,2,4,8,12,24,48 hours after dosing
Population: 24 participants were enrolled; however, the data for the four 2-5 years old participants were not analyzed.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | 6-12 Years of Age Olmesartan Group | 13-16 Years of Age Olmesartan Group
Number analyzed (Participants) | 10 | 10
L/hr | 0.090 (0.029) | 0.079 (0.016)

4. Primary Outcome: For Olmesartan, the Maximum Plasma Concentration Over the Entire Sampling Phase
Time Frame: PK samples were collected pre-dose and at 1,2,4,8,12,24,48 hours after dosing
Population: 24 participants were enrolled; however, the data for the four 2-5 years old participants were not analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 6-12 Years of Age Olmesartan Group | 13-16 Years of Age Olmesartan Group
Number analyzed (Participants) | 10 | 10
ng/mL | 1227 (451) | 895 (262)

5. Primary Outcome: Foe Olmesartan, the Time of Maximum Plasma Concentration
Time Frame: PK samples were collected pre-dose and at 1,2,4,8,12,24,48 hours after dosing
Population: 24 participants were enrolled; however, the data for the four 2-5 years old participants were not analyzed.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | 6-12 Years of Age Olmesartan Group | 13-16 Years of Age Olmesartan Group
Number analyzed (Participants) | 10 | 10
hr | 2.8 (1.3) | 2.5 (1.1)

6. Primary Outcome: For Olmesartan, the Elimination Half-life of the Drug in Plasma
Time Frame: PK samples were collected pre-dose and at 1,2,4,8,12,24,48 hours after dosing
Population: 24 participants were enrolled; however, the data for the four 2-5 years old participants were not analyzed.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | 6-12 Years of Age Olmesartan Group | 13-16 Years of Age Olmesartan Group
Number analyzed (Participants) | 10 | 10
hr | 8.4 (2.4) | 9.1 (1.9)

7. Primary Outcome: For Olmesartan, the Apparent Oral Clearance
Time Frame: PK samples were collected pre-dose and at 1,2,4,8,12,24,48 hours after dosing
Population: 24 participants were enrolled; however, the data for the four 2-5 years old participants were not analyzed.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | 6-12 Years of Age Olmesartan Group | 13-16 Years of Age Olmesartan Group
Number analyzed (Participants) | 10 | 10
L/hr | 4.3 (1.9) | 6.1 (2.6)

8. Primary Outcome: For Olmesartan, the Apparent Oral Volume of Distribution
Time Frame: PK samples were collected pre-dose and at 1,2,4,8,12,24,48 hours after dosing
Population: 24 participants were enrolled; however, the data for the four 2-5 years old participants were not analyzed.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 6-12 Years of Age Olmesartan Group | 13-16 Years of Age Olmesartan Group
Number analyzed (Participants) | 10 | 10
L | 50.9 (20.7) | 81.3 (42.1)

ADVERSE EVENTS:
Time Frame: <3 days
Description: Adverse events observed by the Investigator, or reported by the subject, and any remedial action taken, were recorded in the CRF by the Investigator. The nature of each event, time of onset after drug administration, duration, and intensity were documented together with the Investigator's opinion of the causal relationship to the treatment.
Arm/Group | Olmesartan Group - 2 to 5 Years Old | Olmesartan Group - 6 to 12 Years Old | Olmesartan Group - 13 to 16 Years Old
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/4 | 2/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan Group - 2 to 5 Years Old (N=4) | Olmesartan Group - 6 to 12 Years Old (N=10) | Olmesartan Group - 13 to 16 Years Old (N=10)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Abnormal urine analysis (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No